CLINICAL TRIAL: NCT01133509
Title: A Model for the Implementation of the Cervical Cancer Screening and HPV Vaccination in the Emergency Department: a Pilot Study.
Brief Title: A Model for Implementation of Cervical Cancer Screening and HPV Vaccination the Emergency Department: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alicia Devine, MD, Principal Investigator, Eastern Virginia Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33249
Record Dates: First submitted 2008-11-04; First posted 2010-05-31 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Genital Human Papilloma Virus Infection
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gardisil (Other): gardisil
  Interventions: Drug: Gardasil

INTERVENTIONS:
Drug: Gardasil — 0.5ml IM for three doses, Second and third dose to be given at 2 months and 6 months
  Other Names: Human Papillomarvirus, HPV vaccine, Gardisil, Silgard

SUMMARY:
In this pilot study, we intend to demonstrate that a great portion of women at high risk (inadequate screening, HPV 16/18 and/or cytology) are presenting to the ED, cytology/ HPV testing via ThinPrep®Pap testTM and surveillance. We intend to provide improved access to healthcare and monitoring through administration of vaccine to eligible patients and 1 year follow up for patients involved in this study.

Females meeting inclusion/exclusion criteria participating in the study (n=100) that have not had a cytology test in 2 or more years will be offered the Thin Prep® cytology test. This study will allow surveillance of disease through cytology and HPV DNA testing via collection of data using Thin Prep® cytology with reflex HPV DNA testing according to established guidelines as described below.

Provide improved access to healthcare and monitoring through administration of vaccine for eligible females as established by guidelines. Patients will receive first vaccine in the ED and will have arranged follow up for administration of the 2 month and 6 month series of the HPV vaccination. Through data collection, we intend to determine if there is a need for vaccination and determine if patients are likely to follow up..

ELIGIBILITY:
Inclusion Criteria:

* 3 years of beginning sexual activity or by age 21 years whichever occur first.
* resident of the City of Norfolk, Virginia
* uninsured

Exclusion Criteria:

* Pregnant women
* Women with Hysterectomy with cervical excision
* Women who received full HPV vaccine series
* Known history of cervical cancer
* Male sex
* Loop electrocautery excision procedure(LEEP)
* Cold-Knife conization

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that a great portion of women at high risk (inadequate screening, HPV 16/18 and /or cytology)are presenting to the ED,by analysis of a constructed survey,cytology/HPV testing via ThinPrep Pap test and surveillance | two years

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Devine, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

REFERENCES:
- [Background] Bosch X, Harper D. Prevention strategies of cervical cancer in the HPV vaccine era. Gynecol Oncol. 2006 Oct;103(1):21-4. doi: 10.1016/j.ygyno.2006.07.019. Epub 2006 Aug 17. No abstract available. PMID 16919714
- [Background] Lonky NM. Risk factors related to the development and mortality from invasive cervical cancer clinical utility and impact on prevention. Obstet Gynecol Clin North Am. 2002 Dec;29(4):817-42, viii. doi: 10.1016/s0889-8545(02)00021-9. PMID 12509097
- [Background] Society of Gynecologic Oncologists Education Resource Panel Writing group; Collins Y, Einstein MH, Gostout BS, Herzog TJ, Massad LS, Rader JS, Wright J. Cervical cancer prevention in the era of prophylactic vaccines: a preview for gynecologic oncologists. Gynecol Oncol. 2006 Sep;102(3):552-62. doi: 10.1016/j.ygyno.2006.07.022. PMID 16979432
- [Background] Kinney W, Sung HY, Kearney KA, Miller M, Sawaya G, Hiatt RA. Missed opportunities for cervical cancer screening of HMO members developing invasive cervical cancer (ICC). Gynecol Oncol. 1998 Dec;71(3):428-30. doi: 10.1006/gyno.1998.5135. PMID 9887244
- [Background] Plummer M, Schiffman M, Castle PE, Maucort-Boulch D, Wheeler CM; ALTS Group. A 2-year prospective study of human papillomavirus persistence among women with a cytological diagnosis of atypical squamous cells of undetermined significance or low-grade squamous intraepithelial lesion. J Infect Dis. 2007 Jun 1;195(11):1582-9. doi: 10.1086/516784. Epub 2007 Apr 16. PMID 17471427
- See also: American Cancer Society — http://www.cancer.org/docroot/home/index.asp?level=0
- See also: American College of Obstetrics and Gynecology — http://www.acog.org/
- See also: United States Preventative Service Task Force — http://www.ahrq.gov/clinic/uspstfix.htm